CLINICAL TRIAL: NCT06177717
Title: The American Lung Association (ALA) Deep Phenotyping Ancillary Study of the Lung Health Cohort (LHC)
Brief Title: Deep Functional Phenotyping of the ALA Lung Health Cohort
Acronym: DLP-LHC
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); American Lung Association (Other); University of Vermont (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00273188; U01HL146408-01 (NIH)
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about lung structure and function in a group of 1000 healthy people aged 25 to 35. The main questions it aims to answer are whether people's bodies, environment, and general lung health are associated with:

* the structure of the participants lungs' airways,
* the structure of blood vessels in the participants lungs and heart, and
* the participants lungs' ability to exchange gases.

Participants will take four different lung function tests to measure lung function, including:

* air movement in the lungs (oscillometry)
* lung size (slow vital capacity (SVC) and functional residual capacity (FRC)
* gas transfer in the lungs (diffusing capacity for carbon monoxide (DLCO).

DETAILED DESCRIPTION:
The parent Lung Health Cohort (LHC) study will leverage the national infrastructure of the American Lung Association's (ALA) Airways Clinical Research Centers (ACRC) to form the first national cohort of adults focused on respiratory health. The parent LHC study will recruit approximately 4000 community-dwelling adults aged 25-35 from metropolitan regions across the U.S. for the purpose of defining lung health and developing targets to intercept chronic lung disease at its earliest stages.

The parent LHC study will be examining a multitude of known and potential factors related to reduced reserve and increased susceptibility to lung disease, such as childhood and adult health status, infections and exposures. Two of the primary outcomes being assessed during this cross-sectional phase of the parent LHC will be spirometry, measured in forced expiratory volume in 1 second (FEV1), respiratory symptoms in relation to environmental exposures, measured in exposure to particulate matter under 2.5 microns in size (PM2.5). These will be assessed in relation to computed tomography (CT) measures of lung injury. The ancillary study expands the phenotyping to include detailed measurements of lung structure and function, including lung volumes, oscillometry, diffusing capacity for carbon monoxide (DLCO), and airway, blood vessel and cardiac morphology by CT. This deeper phenotyping will move the characterization of lung health reserve beyond FEV1, as well as establish a more comprehensive baseline of lung health to allow assessment of susceptibility. Furthermore, the investigators will relate these detailed measures of lung structure and function to modifiable exposures and risk factors that will allow identification of risks to lung health and potential strategies to mitigate risk. The investigators hypothesize that modifiable exposures and risk factors influence lung health by the effects on structural and functional dysanapsis of the airway, parenchyma and pulmonary vasculature, as well as cardiac morphology and gas exchange.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-35 years at the time of the baseline examination
* Able to read and understand English or Spanish
* Has a social security number
* Resident (citizen or non-citizen) of the United States (US) for at least 12 months prior to examination.

Note: Individuals who are residents of the US who have temporarily spent time living outside of the US during the last 12 months (e.g., student exchange program, military posting) are eligible for participation.

* Willing to provide contact information for at least 2 proxies who are likely to know the whereabouts and vital status of the participant

Exclusion Criteria:

1. Severe asthma, which is defined as any of the following:

   * Current (i.e. at the time of the visit) Global Initiative for Asthma (GINA) Step 4 or higher therapy (medium dose inhaled corticosteroid/long-acting beta agonist (ICS/LABA) or high dose inhaled corticosteroid [ICS] or add-on long-acting muscarinic antagonist (LAMA); Medium dose = >250 fluticasone, propionate =100 fluticasone furoate, >200 beclomethasone, >400 budesonide, >220 mometasone). The investigators will accept low-dose ICS/LABA or medium dose ICS.

   OR
   * 3 or more unscheduled healthcare visits (provider/urgent care/ER) for asthma in the past 12 months OR
   * One asthma hospitalization in the past 12 months
2. History of any chronic lung disease other than asthma including but not limited to chronic obstructive pulmonary disease (COPD), cystic fibrosis, pulmonary fibrosis, pulmonary hypertension
3. Current pregnancy
4. History of cancer other than non-melanoma skin cancer
5. Diagnosed cardiovascular diseases (i.e., congenital heart disease, coronary heart disease)
6. Inability to comply with study procedures, including

   * Inability or unwillingness to provide informed consent
   * Inability to perform study measurements
   * Inability to be contacted by phone (via calls and/or text messaging) or email
7. Any condition in the opinion of the physician that puts the participant at risk by participating in the study (e.g., serious respiratory illness requiring antibiotics or steroids or severe fever at the time of the study visit).
8. Institutionalization

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young adults between 25 and 35 years of age at baseline
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Associations with airway-parenchymal dysanapsis | Baseline
  Correlation of adverse modifiable exposures and risk factors with increased airway-parenchymal dysanapsis
Associations with vascular parenchymal dysanapsis and cardiac chamber size | Baseline
  Correlation of adverse modifiable exposures and risk factors with increased vascular parenchymal dysanapsis and increased cardiac chamber size
Associations with diffusing capacity for carbon monoxide (DLCO) | Baseline
  Correlation of adverse modifiable exposures and risk factors with lower diffusing capacity for carbon monoxide (DLCO)

CONTACTS AND LOCATIONS:
Overall Officials: Meredith McCormack, MD, Principal Investigator — Johns Hopkins University
Locations (12):
- United States (12):
  - University of Alabama, Birmingham, Alabama
  - University of California, Los Angeles, Los Angeles, California
  - National Jewish Health, Denver, Colorado
  - Nemours Children's Jacksonville, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - University of Kansas, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Duke University, Durham, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - University of Pittsburgh - Emphysema/COPD Research Center, Pittsburgh, Pennsylvania
  - University of Vermont, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Yes
Deidentified study data will be made available to researchers by publishing on a data sharing site. Data will be made available upon completion of the study and publication of the summary paper.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made available indefinitely upon completion of the study (anticipated 6/30/2028).